CLINICAL TRIAL: NCT00446654
Title: A Phase Ib Randomized Open Label Study Between Once-every-two-weeks and Once-every-four-weeks Treatment of CGC-11047 in Patients With CNV Due to Age Related Macular Degeneration
Brief Title: Safety of 16.5 mg (3.3%) CGC-11047 Once Every 2 Weeks vs. Once Every 4 Weeks in Patients With CNV Due to AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47-MD-002
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-06

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — CGC 11047; (N(1),N(12))bis(ethyl)-6,7-dehydrospermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGC-11047 once every 2 weeks (Experimental): 16.5 mg CGC-11047 as a subconjunctival injection once every two weeks.
  Interventions: Drug: CGC-11047
- CGC-11047 once every four weeks (Experimental): 16.5 mg CGC-11047 as a subconjunctival injection once every four weeks.
  Interventions: Drug: CGC-11047

INTERVENTIONS:
Drug: CGC-11047 — 16.5 mg (3.3%) subconjunctival injection
  Other Names: PG11047

SUMMARY:
The purpose of this research study is to determine how safe and effective subconjunctival injections of CGC-11047 are in subjects with wet age related macular degeneration at two different dosing intervals.

DETAILED DESCRIPTION:
The purpose of this research study is to determine how safe and effective subconjunctival injections of CGC-11047 are in subjects with wet age related macular degeneration at two different dosing intervals. Half of the participants in the study will receive CGC-11047 every two weeks and half of the participants in the study will receive CGC-11047 every four weeks. If your doctor determines that you are eligible for the study based on his/her judgement and according to the entry requirements set by the sponsor of the research, you will be randomly assigned (by chance, like the flip of a coin), to receive CGC-11047 every two weeks or every four weeks. Whether you receive drug every two weeks or every four weeks, you will still need to come to the clinic approximately every two weeks for the first three months, and approximately four times after that until it has been at least 12 months since you received your first treatment of study drug.

Two studies (this one and another one) are occurring to test CGC-11047 in patients with wet age-related macular degeneration for the first time. However, this drug (CGC-11047) is being studied in cancer patients at doses much higher than will be given to any subjects in either of these studies. The cancer patients have tolerated the drug well with the exception of one cancer patient who had two reactions to the drug (pancreatitis and hypotension). However, this patient had advanced cancer (non-Hodgkin's lymphoma with a life expectancy of less than 3 months) and received 38X the dose to be administered in this AMD study. Aside from this one patient, there have not been any serious side effects related to the drug.

This study will involve about 100 subjects at about 15 different sites internationally.

The study will take place over 12 months and will include about 12 office visits to the study doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of subfoveal choroidal neovascularization secondary to AMD in the study eye, with leaking present on a fluorescein angiogram as determined by the clinical investigator.
2. Visual acuity: BCVA in the study eye between 20/40 and 20/320 and better than or equal to 20/320 in the fellow eye.
3. Patients who refuse standard of care or have not benefited from standard of care in the opinion of the principal investigator.
4. Clear ocular media and adequate pupillary dilatation to permit good quality ophthalmologic exam.
5. Male or female patients aged >= 50 years.
6. Ability to understand and the willingness to sign a written informed consent document and return for all study visits.

Exclusion Criteria:

1. Patients with CNV not due to AMD in the study eye.
2. Patients with a retinal tear in the study eye.
3. Patient has a subretinal hemorrhage that comprises more than 50% of total lesion size, or has atrophy or fibrosis in the center of fovea.
4. Patients who have undergone intraocular surgery within 2 months or extrafoveal/juxtafoveal laser within 3 months of study entry in the study eye.
5. Any macular disease other than AMD causing vision loss in either eye.
6. Active infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye. Anterior segment diseases such as blepharitis, ocular rosacea, lid problems which could increase the risk of infection after study drug injection.
7. Uncontrolled glaucoma (defined as intraocular pressure >25 mmHg (P0) on maximum medical therapy) or clinically significant glaucomatous visual field loss in both eyes.
8. Significant media opacities, including cataract that might interfere with visual acuity, assessment of toxicities or fundus photography in the study eye in the judgement of the clinical investigator.
9. Spherical refractive error more than -8.0 diopters in the study eye.
10. Use of any approved or investigational AMD agent (standard of care) within four weeks of study enrollment.
11. Use of any systemic investigational agent within 30 days of study enrollment.
12. Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patients with a clinically significant or symptomatic cardiac arrhythmia, recent myocardial infarction (within 6 months), or evidence of a current significant ventricular conduction abnormality.
14. Women who are pregnant or breast-feeding.
15. Women of childbearing potential and male patients who are partners of women of childbearing potential who are unwilling to use approved, effective means of contraception according to the institution's standards.
16. Allergy to fluorescein dye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — Wilmer Eye Institute, Johns Hopkins Hospital School of Medicine
Locations (8):
- Wilmer Eye Institute, Baltimore, Maryland, United States
- Dr. Quiroz-Mercado, Mexico City, District Federal, Mexico
- Russia (6):
  - Federal State Establishment "Intersectoral Research and Technology Complex "Eye Microsurgery" named by Academic SN Fyodorov of Federal Agency for Healthcare and Social Development, Cheboksary
  - Federal State Establishment "Intersectoral Research and Technology Complex "Eye Microsurgery" named by Academic SN Fyodorov of Federal Agency for Healthcare and Social Development, Moscow
  - Closed Joint Stock Company "Inter YuNA", Rostov-on-Don
  - Federal State Establishment "Intersectoral Research and Technology Complex "Eye Microsurgery" named by Academic SN Fyodorov of Federal Agency for Healthcare and Social Development, Saint Petersburg
  - Saint Petersburg State Healthcare Establishment "City Consultative Diagnostic Centre #1", Saint Petersburg
  - State Educational Establishment of Higher Professional Education "Military Medical Academy named by SM Kirov", Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period spanned 05 February 2007 to 10 July 2007. Patients were randomised to one of the two treatment groups. Treatment group assignment for each patient was made centrally.
Period: Overall Study
Arm/Group | CGC-11047 Once Every 2 Weeks | CGC-11047 Once Every Four Weeks
Started | 21 | 22
Completed | 19 | 22
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGC-11047 Once Every 2 Weeks | CGC-11047 Once Every Four Weeks | Total
Number analyzed (Participants) | 21 | 22 | 43
Age Categorical [Number; unit: participants] — Demographic data is missing for 5 patients.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 7 | 3 | 10
    >=65 years | 13 | 15 | 28
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data is missing for 5 patients.
  years | 69.3 (8.5) | 68.1 (7.0) | 68.7 (7.7)
Gender [Number; unit: participants] — Demographic data is missing for 5 patients.
  participants
    Female | 12 | 12 | 24
    Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
  Mexico | 5 | 1 | 6
  Russian Federation | 14 | 20 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Safety of 2-weekly or 4-weekly Administration of CGC-11047
Time Frame: 3 months
Reporting Status: Not Posted

2. Secondary Outcome: To Evaluate Possible Suppression and/or Regression of Choroidal Neovascularization
Time Frame: 3 months
Reporting Status: Not Posted

3. Primary Outcome: Change in Baseline to 3 Months in Best Corrected Visual Acuity
Description: Visual acuity was measured with a standard eye exam using the preferred research based eye chart (LogMar chart). On the LogMar chart each letter has a score value of 0.02 log units. LogMAR VA = 0.1 + LogMAR value of the best line read - 0.02 X (number of letters read).
  The outcome measure presented is the difference in LogMAR between baseline and at three months.
Time Frame: Baseline and 3 months
Population: Analysis was performed on all patients who received at least one treatment.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CGC-11047 Once Every 2 Weeks | CGC-11047 Once Every Four Weeks
Number analyzed (Participants) | 21 | 21
logMAR | -0.01 (0.21) | 0.08 (0.25)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CGC-11047 Once Every 2 Weeks | CGC-11047 Once Every Four Weeks
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/22
Other Adverse Events (participants affected / at risk) | 7/21 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGC-11047 Once Every 2 Weeks (N=21) | CGC-11047 Once Every Four Weeks (N=22)
Strangulate umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of visual acuity (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGC-11047 Once Every 2 Weeks (N=21) | CGC-11047 Once Every Four Weeks (N=22)
Conjunctival haemorrhage (Eye disorders) | 2 (4) | 1 (1)
Eye pain (Eye disorders) | 6 (12) | 1 (1)
Foreign body sensation in eye (Eye disorders) | 2 (5) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 1 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed: 100 patients were planned; 43 patients were recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No